CLINICAL TRIAL: NCT03925311
Title: Transcriptome Profiling and Immune/ Biochemical Markers of Peripheral Blood to Predict Endometrial Receptivity and Successful Implantation
Brief Title: Transcriptome Profiling and Endometrial Receptivity
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2014.637
Record Dates: First submitted 2019-04-03; First posted 2019-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
Keywords: Transcriptome; endometrial receptivity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endometrial biopsy and blood sampling — patient will be performed endometrial biopsy and collected blood samples at particular time points

SUMMARY:
The aim of this study is to correlate and identify the biochemical markers which may reflect WOI. Blood samples will be collected and endometrial biopsy will be performed at particular time points.

DETAILED DESCRIPTION:
Endometrial receptivity in the midluteal phase of the menstrual cycle, known as the window of implantation (WOI), occurs only for a very short period of time. However, so far, there is no reliable clinical and biochemical indicators of WOI. Therefore, this study is to correlate and identify the biochemical markers which may reflect WOI.

participants will be asked to be:

1. performed endometrial biopsy
2. taken blood for a few time points (e.g. pre-conception and being pregnant) and to compare different kinds of biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

Age 20-40 years.

Exclusion Criteria:

* Uncorrected uterine anomalies, such as septate or bicornuate uterus, fibroids (submucous/intramural).
* Intrauterine adhesions.
* Adenomyosis.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — This study only focuses on female group
Study Population: Subjects will be recruited from the Prince of Wales Hospital.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2015-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of the transcriptome profiling in the peripheral blood | From the day of endometrial biopsy through study completion, an average of 2 months
  RNA per sample will be prepared into two portions. One is for RNA sequencing and the other is for small RNA sequencing. The next step is hydrolysis of RNA into 200-300 nucleotides prior to reverse transcription. When sequencing RNA other than mRNA the library preparation is modified. The cellular RNA is selected based on the desired size range. For miRNA, the RNA is isolated through size selection. Once isolated, linkers are added to the 3' and 5' end then purified. The final step is cDNA generation through reverse transcription.
The change of the immune markers in the peripheral blood | From the day of endometrial biopsy through study completion, an average of 2 months
  Immune markers including cytokines such as leukemia inhibitory factor, macrophage colony stimulating factor, interleukin - 1 beta, transforming growth factor beta-1, Tim-3, galectin-9 and other markers considered to play a role in implantation will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided